CLINICAL TRIAL: NCT06155305
Title: Consistency of Organoids Based Drug Sensitivity and Efficacy of Neoadjuvant Chemotherapy in Breast Cancer
Brief Title: Organoids Based Drug Sensitivity in Neoadjuvant Chemotherapy of Breast Cancer
Acronym: ONAC
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0840
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Organoids; Breast Cancer; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The primary tumor tissue and blood will be stored and used to identify potential biomarker for chemotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients: Patients diagnosed with breast cancer undergo biopsy before initiating neoadjuvant therapy.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Before initiating neoadjuvant therapy, patients diagnosed with breast cancer undergo a tumor biopsy. The tissue obtained from the biopsy is utilized to establish organoids and conduct drug testing.

SUMMARY:
Breast cancer is the most common malignancy in women worldwide. Patients with breast cancer are often diagnosed at later stages and have a strong desire for breast conservation, necessitating neoadjuvant chemotherapy. Tumors of different molecular subtypes and individual variations among patients lead to significant differences in treatment efficacy. Precise assessment of patients' responses to treatment regimens is imperative in advancing prognosis of breast cancer. In this study, 58 patients diagnosed with breast cancer and scheduled for neoadjuvant therapy will be recruited. Patient-derived organoids from their tumor biopsies will be utilized to evaluate the sensitivity of chemotherapy regimen. These drugs primarily include Doxorubicin, Carboplatin, Cyclophosphamide, Paclitaxel, as well as targeted therapies such as Herceptin and Pertuzumab.

DETAILED DESCRIPTION:
58 early-stage breast cancer patients scheduled to undergo neoadjuvant therapy will be recruited. Baseline information including medical history, ultrasound, Breast-Specific Gamma Imaging (BSGI), and magnetic resonance imaging (MRI) records, will be collected both before and after two cycles of chemotherapy. Tumor tissue from these patients will be obtained via biopsies guided by ultrasound. Patient-derived organoids (PDOs) will be established and cultured from the collected tumor tissue. Subsequently, these PDOs will be subjected to treatment with drugs from standard chemotherapeutic regimens for breast cancer. The growth of the organoids will be assessed post-treatment, and dose-response curves will be generated. For evaluating the clinical outcomes of the patients, the Residual Cancer Burden (RCB) system will be used to evaluate tumor histological responses in patients. The consistency between treatment responses observed in the PDO models and the clinical outcomes of patients will be evaluated through correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form and willingness to participate in the clinical study.
2. Female patients aged between 18 and 70 years old.
3. Confirmed early-stage breast cancer eligible for surgery (AJCC stages I to IIIA), with a tumor diameter of ≥ 2cm detected by MRI and without distant metastasis (M0).

   The largest lesion among multiple lesions has a diameter of ≥ 2cm.
4. ECOG performance status score of 0-1.
5. No significant abnormalities in liver and kidney function (BIL <1.5-fold upper limit of normal (ULN)；ALT<2.5×ULN; AST<2.5×ULN；Crea≤1×ULN).

Exclusion Criteria:

1. Received prior treatments.
2. Locally advanced breast cancer not amenable to surgery or inflammatory breast cancer (AJCC stage unresectable III).
3. Bilateral breast cancer.
4. Multiple breast cancers distributed in different quadrants.
5. Patients not suitable for neoadjuvant chemotherapy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male breast cancer is a rare disease.
Study Population: Patients with breast cancer (AJCC stages I to IIIA) who need to receive neoadjuvant therapy.
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between drug sensitivity test results in patient-derived organoid models and clinical outcomes. | 2023.12-2025.06
  The drug sensitivity test results obtained from patient-derived organoid models will be compared with the clinical outcomes.

SECONDARY OUTCOMES:
Comparison between drug sensitivity of organoid models and clinical imaging (MRI, ultrasound, BSGI) in predicting the efficacy of neoadjuvant chemotherapy. | 2023.12-2025.06
  The sensitivity and specificity would be checked between drug sensitivity of organoid models and clinical imaging (MRI, ultrasound, BSGI) in predicting the efficacy of neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, Principal Investigator — 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Zhigang Chen, Principal Investigator — 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China